CLINICAL TRIAL: NCT02226458
Title: An Exploratory Open-Label Phase 2 Study of EPI-743 (Vincerinone TM) in Children With Autism Spectrum Disorder
Brief Title: An Exploratory Open Label Study of EPI-743 (Vincerinone TM) in Children With Autism Spectrum Disorder
Acronym: Autism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was halted prior to enrolling.
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI743-14-025
Record Dates: First submitted 2014-08-21; First posted 2014-08-27 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Mitochondrial Disorders; EPI-743; EPI743; Rett syndrome; Angelman syndrome
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Mitochondrial Diseases; Rett Syndrome; Angelman Syndrome | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-743 (Experimental): 15 mg/kg oral solution three times per day, maximum of 200 mg per dose
  Interventions: Drug: EPI-743

INTERVENTIONS:
Drug: EPI-743
  Other Names: Vincerinone TM

SUMMARY:
The investigators hypothesize that EPI-743 may provide clinical benefit to children with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
An Exploratory Open Label Phase 2 Study of EPI-743 (Vincerinone TM) in Children with Autism Spectrum Disorder

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Autism Spectrum Disorder as defined by the DSM-V criteria for ASD and a gold-standard diagnostic evaluation for ASD such as the Autism Diagnostic Observation Schedule (ADOS) and/or the Autism Diagnostic Interview - Revised (ADI-R)
2. Male or female, 3 years to 14 years of age
3. Abnormal glutathione cycle biomarkers (GSH/GSSG in plasma<8.0)
4. Language impairment (as defined by the CELF-2 or CELF-4 screener)
5. Ability to complete language assessment (using either CELF or PLS)
6. Subject or subject's guardian able to consent and comply with protocol requirements
7. Abstention from use of Coenzyme Q10, vitamin E, lipoic acid, folinic acid, other forms of folic acid above recommended daily allowance (RDA), and idebenone 2 months prior to treatment with EPI-743 and for duration of study
8. Stable regimen of medication and supplements for 2 months prior to enrollment and duration of the study

Exclusion Criteria:

1. Allergy to EPI-743 or sesame oil
2. Allergy to vitamin E
3. Clinical history of bleeding or abnormal baseline PT/PTT
4. Use of anticoagulant medications
5. Participation in any other interventional study within 90 days of treatment.
6. Use of antipsychotic medications
7. Moderate to severe positive response on ABC irritability subscale on questions: Injures self on purpose, is aggressive to other children or adults (verbally or physically), deliberately hurts himself/ herself, and/or does physical violence to self
8. Severe impairment as defined as a Vineland Adaptive Behavioral Scales composite standard score of <40
9. Patients with genetic disease that gives rise to ASD (e.g. Rett syndrome, Down syndrome, fragile x syndrome)
10. Abnormal liver function tests two times the upper limit of normal or renal insufficiency with creatinine levels two times the upper limit of normal

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-11-30 (Estimated); Study Completion 2016-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy | 6 months
  Change in plasma levels of reduced and oxidized glutathione from baseline to six months

SECONDARY OUTCOMES:
Secondary Endpoint | 6 months
  Change in language skills as assessed by change from baseline to six months on the Clinical Evaluation of Language Fundamentals or Preschool Language Scale
Secondary Endpoint | 6 months
  Change from baseline to six months in adaptive behavior and social skills as assessed by the Vineland Adaptive Behavior Scale-Second Edition (VABS), Social Responsiveness Scale (SRS), and computerized eye movement analysis
Secondary Endpoint | 6 months
  Change from baseline to six months in stereotyped behavior and associated ASD symptoms as assessed by Aberrant Behavior Checklist (ABC), The Ohio Autism Clinical Impression Scale (OACIS), Repetitive Behavior Scale - Revised (RBS-R) and Autism symptoms questionnaire (ASQ)
Secondary Endpoint | 6 months
  Change from baseline to six months in gastrointestinal function as assessed by Symptom Diary (stool frequency, abdominal symptoms and medications) and six-item GI severity index (6-GSI).
Secondary Endpoint | 6 months
  Change from baseline to six months in caregiver strain experienced by parents of children with emotional and behavioral disorders as assessed by Caregiver Strain Questionnaire (CGSQ)
Secondary Endpoint | 6 months
  Change from baseline to six months in intellectual function, attention and memory as assessed by Leiter-R test
Secondary Endpoint | 6 months
  Change from baseline to six months in biomarkers of oxidative stress
Secondary Endpoint | 6 months
  Pharmacokinetic Assessment of EPI-743 including maximal plasma concentration (Cmax), area under plasma concentration curve (AUC), apparent oral clearance, apparent volume of distribution and time to peak concentration
Safety Endpoint | 8 months
  To examine the safety of EPI-743 in subjects with Autism Spectrum Disorder by examining drug-related adverse and serious adverse events